CLINICAL TRIAL: NCT02203227
Title: Efficacy and Safety Study of Dietary Supplements (BioTurmin, BioTurmin-WD and MaQxan) on Cotinine Level and Oxidative Stress Marker in Chronic Smokers Having Mild to Moderate Hyperlipidemia
Brief Title: Efficacy and Safety Study of Dietary Supplements in Chronic Smokers Having Mild to Moderate Hyperlipidemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Olive Lifesciences Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OLS-SH/06-14 VER 01
Record Dates: First submitted 2014-07-28; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Smokers; Hyperlipidemia
Keywords: Dietary supplements; Cotinine level; Malondialdehyde; Chronic smokers; Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Capsule containing 250 mg of placebo, two times a day
  Interventions: Dietary Supplement: Placebo
- BioTurmin (Experimental): Capsule containing 250 mg of BioTurmin (Curcuma longa rhizomes extract), two times a day
  Interventions: Dietary Supplement: BioTurmin (Curcuma longa rhizomes extract)
- BioTurmin-WD (Experimental): Capsule containing 250 mg of BioTurmin-WD (water dispersible curcuminoids), two times a day
  Interventions: Dietary Supplement: BioTurmin-WD (Water dispersible curcuminoids)
- MaQxan (Experimental): Capsule containing 10 mg of MaQxan (Tagetes erecta flower extract), two times a day
  Interventions: Dietary Supplement: MaQxan

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: Placebo
Dietary Supplement: BioTurmin (Curcuma longa rhizomes extract)
  Arms: BioTurmin
Dietary Supplement: BioTurmin-WD (Water dispersible curcuminoids)
  Arms: BioTurmin-WD
Dietary Supplement: MaQxan
  Arms: MaQxan

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of dietary supplements (BioTurmin, BioTurmin-WD and MaQxan) on cotinine level and oxidative stress marker in chronic smokers having mild to moderate hyperlipidemia after 30 and 60 days of intervention.

DETAILED DESCRIPTION:
In a randomized, double-blind, placebo control trial, the efficacy and safety of dietary supplements (BioTurmin, BioTurmin-WD and MaQxan) will be investigated in chronic smokers having mild to moderate hyperlipidemia. Sixty subjects will be randomly assigned to receive the dietary supplements and placebo for 60 days. The efficacy of the supplements will be measured by estimating cotinine and malondialdehyde level.

ELIGIBILITY:
Inclusion Criteria:

* Men > 20 years
* Chronic cigarette/ beedi smoker (2-3 packets/day since last 3 years or more) with mild to moderate hyperlipidemia (LDL ranging 160-189 mg/dL, TC >200 mg/dL and/or HDL-C <40 mg/dL)
* Being mentally competent and able to understand all study requirements and sign the informed consent form.

Exclusion Criteria:

* Patients with Chronic obstructive pulmonary disease (COPD)
* Women
* Patients with severe liver, renal, cardiac or brain diseases.
* Unable to complete follow up.
* Subjects on any medication like diuretics.
* Allergic to any medication.
* With a history of alcohol and/or drug abuse.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
change in urine cotinine and serum oxidative stress marker (malondialdehyde) level | Baseline, on day 30 and on day 60

SECONDARY OUTCOMES:
Change in serum lipid profile | Baseline, on day 30 and on day 60
  Low density lipoprotein-cholesterol (LDL-C), very low density lipoprotein-cholesterol (VLDL-C), high density lipoprotein-cholesterol (HDL-C), total cholesterol (TC)

OTHER OUTCOMES:
Safety and tolerability (composite measure) | Baseline, on day 30 and on day 60
  Physical and clinical laboratory evaluations - Electrocardiogram (ECG), haematology [complete blood count (CBC)], biochemical tests (serum urea, serum creatinine), liver function test and urine analysis

CONTACTS AND LOCATIONS:
Overall Officials: Venkateshwarlu K, MD (Ayur), Principal Investigator — Sreenivasa Clinic Diabetic Research Center
Locations (1):
- Sreenivasa Clinic Diabetic Research Center, Bangalore, Karnataka, India

REFERENCES:
- See also: Dietary supplements — http://www.nlm.nih.gov/medlineplus/dietarysupplements.html
- See also: Curcuma longa — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0977052440&QV1=CURCUMA+LONGA
- See also: Tagetes erecta — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0090131434&QV1=TAGETES+ERECTA+EXTRACT